CLINICAL TRIAL: NCT03603405
Title: Phase I-II Study Evaluating HSV-tK + VALACYCLOVIR GENE THERAPY Combination with Radiotherapy and Chemotherapy for Newly Diagnosed Anaplastic Astrocytoma and Glioblastoma Multiforme.
Brief Title: HSV-tk and XRT and Chemotherapy for Newly Diagnosed GBM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, David Baskin MD, Sponsor-Investigator and Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018178
Record Dates: First submitted 2018-07-01; First posted 2018-07-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma
Keywords: GBM, AA, Glioblastoma, Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Genetic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: ADV/HSV-tk (gene therapy) (Experimental): Experimental: ADV/HSV-tk (gene therapy)
  The gene therapy investigational product, HSV-tk will be injected during the surgery. Within 24 hours valacyclovir will be given for 14 days. Radiotherapy will be administered over 30 sessions (over 6 weeks) starting within 9 days of surgery. Standard of care/routine chemotherapy will be started concurrent with the radiotherapy dependent on patient status based on best clinical judgment following the Stupp protocol.
  Patient can receive second treatment of HSV-tk after 6 months.
  Interventions: Drug: ADV/HSV-tk (gene therapy)

INTERVENTIONS:
Drug: ADV/HSV-tk (gene therapy) — The investigational adenovirus gene therapy injected at tumor site followed by valacyclovir, radiotherapy, and chemotherapy
  Other Names: gene therapy, gene therapy; HSV-tk

SUMMARY:
Study to assess the safety and efficacy of HSV-tk (gene therapy), valacyclovir, radiotherapy and chemotherapy in newly diagnosed glioblastoma multiforme (GBM) or anaplastic astrocytoma (AA).

DETAILED DESCRIPTION:
This is a prospective, phase I-II study to assess the efficacy and toxicity of HSV-tk + valacyclovir gene therapy in combination with radiotherapy and standard of care chemotherapy for anaplastic astrocytoma (AA) or glioblastoma multiforme (GBM). This study is comprised of newly diagnosed patients with AA or GBM.

Clinical response will be evaluated by neurological evaluation, neuropsychological testing, and imaging studies as well as by histological examination. Blood samples will be taken for systemic immunological response, blood counts, and liver functions tests. Genetic testing of tumor tissue will be performed, including genetic analysis and cell cultures. Toxicity will be graded by the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 and Radiation Therapy Oncology Group (RTOG) neuro-toxicity scores (see Appendices). Patients will also be followed to assess median time to progression and median survival.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have frozen section biopsy proven anaplastic astrocytoma or glioblastoma multiforme without evidence of multifocal disease defined as multiple lesions greater than 2 cm separate from the primary treatment target, or brainstem involvement as well as radiographic evidence consistent with these diagnoses.
* Life expectancy ≥ 12 weeks.

  - Patient can receive second treatment of HSV-tk after 6 months
* Patients should have the following characteristics: newly diagnosed anaplastic astrocytoma or glioblastoma demonstrated by frozen section biopsy, prior surgery which demonstrated anaplastic astrocytoma or glioblastoma multiforme which requires repeat surgery for residual tumor, but no radiation or chemotherapy has been received, ECOG performance status of 0-1. No evidence of other active malignancy (except squamous or basal cell skin cancers).
* Patients with leptomeningeal disease may be considered for enrollment into the study.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks of the study by the investigator (or his/her designee) with the aid of written information.
* Willing to provide biopsies as required by the study.
* WOCBP must have a negative serum pregnancy test within 7 days prior to the administration of the first study treatment. Women must not be lactating.
* WOCBP and men must practice an effective method of birth control
* Patients must have adequate baseline organ function as assessed by the following laboratory values before initiating the protocol:
* serum creatinine < 1.5 mg/dL
* T. bilirubin < 2.5 mg/dL, ALT, AST, GGT and Alk Phos < 2 x normal
* Platelet count > 100,000/ml , ANC> 1500/ml , Hgb> 10 gm/dL
* Normal partial thromboplastin time (PTT) and Pro-Thrombin Time (PT)

Exclusion Criteria:

* Prior treatment with immunomodulatory therapy, immunotherapy, and/or gene vector therapy in the past 3 months.
* Any cytotoxic chemotherapy, RT, or immunotherapy or any investigational drug within 3 weeks of study treatment start.
* Evidence of substantial multifocal disease defined as multiple lesions greater than 2cm separate from the primary treatment target, or brainstem involvement. Discrete areas of contrast enhancement connected by abnormal T2 FLAIR signal on MRI scan are not considered multifocal disease, as this represents a single tumor.
* Patients with brainstem involvement, in patients with leptomeningeal disease, no evidence of diffuse disease or spread to the spine.
* Patients on immunosuppressive drugs (other than steroids for brain edema).
* In patients with leptomeningeal disease, no evidence of diffuse disease or spread to the spine.
* In patients with leptomeningeal disease, no bulky leptomeningeal metastases with potential to obstruct CSF flow will not be enrolled.
* Liver disease, such as cirrhosis or active/chronic hepatitis B or C.
* History of or current alcohol misuse/abuse within the past 12 months.
* Known or suspected allergy or hypersensitivity to any component of the proposed regimen (gene vector/Valacyclovir).
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications (Valacyclovir).
* No active malignancy except for non-melanoma skin cancer or in situ cervical cancer or treated cancer from which the patient has been continuously disease free for more than 3 years.
* The presence of active CNS toxoplasmosis infection or Progressive Multifocal Leukoencephalopathy demonstrated on CT or MRI imaging
* The presence of active untreated cellulitis or untreated wound infections. Treated and resolving cellulitis and infections are not an exclusion criteria.
* Active IV drug abuse or severe opioid abuse
* Pregnant or breastfeeding women or women/men able to conceive and unwilling to practice an effective method of birth control. WOCBP must have a negative serum pregnancy test within 7 days prior to the administration of the first study treatment.
* Presence of active or suspected acute or chronic uncontrolled infection or history of immunocompromise, including a positive HIV test result.
* Patients < 18 years of age
* Unwilling or unable to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival in months up to 5 years from Study drug administration (Day 0) | Up to 60 months measured in months
  The overall survival rate of patients with Anaplastic Astrocytoma and Glioblastoma in months will be assessed up to 5 years from study drug administration.

SECONDARY OUTCOMES:
Progression free survival assessments will be done every 6-8 weeks for 1st year thereafter every 12-14 weeks until disease progression or death | Up to 60 months measured in months
  Patients will have MRI or CT every 6-8 weeks for the first year post surgery. Thereafter patient will have MRI or CT every 12-14 weeks until completion of the protocol study specific treatment. Progression free survival will be assessed by RANO response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Baskin, MD, Principal Investigator — Houston Methodist Neurological Institute
Locations (1):
- Houston Methodist Neurological Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined